CLINICAL TRIAL: NCT04881071
Title: Randomized Clinical Trial to Evaluate the Efficacy of a Scarf Designed to Facilitate Skin-to-skin Contact Between Parents and Healthy Term Neonates
Brief Title: Efficacy of a Scarf to Facilitate Mother-newborn Contact Designed to Facilitate Skin-to-skin Contact
Acronym: MOKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Consorci Sanitari de l'Alt Penedès i Garraf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CSAPG-14
Record Dates: First submitted 2021-04-30; First posted 2021-05-11 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Full-term Newborn Babies
Keywords: Kangaroo-Mother Care Method

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scarf (Experimental): Two hours after delivery, mothers will be informed of the benefits of the skin-to-skin method, and the towel with which mother and newborn are covered from the moment of delivery will be replaced by a NeoBulleⓇ scarf. This scarf, which can be used by the mother and/or her partner, is specific for practicing the "skin-to-skin" technique. It facilitates breastfeeding posture, keeps the newborn well covered and supported on the back. The NeoBulleⓇ scarf is not a baby carrier device that allows standing or walking without holding the baby with the arms. Nursing staff will ensure the proper understanding of scarf usage instructions by parents and provide them with written instructions. Mother and newborn will remain with the NeoBulleⓇ scarf placed in the delivery area until they are transferred to the hospitalization unit. Once in the hospitalization unit, mothers will have the option to continue contact with the baby using the scarf or dress the newborn.
  Interventions: Device: Scarf
- Usual clinical practice (Active Comparator): Two hours after delivery, mothers will be informed about the benefits of the skin-to-skin method, and the traditional practice in the study centers will be followed, whereby the newborn remains in contact with the mother, covered by a towel, from the moment of birth until both are transferred to the hospitalization unit. In the hospitalization unit, they will have the option to continue in this manner or dress the newborn.
  Interventions: Other: Usual clinical practice

INTERVENTIONS:
Device: Scarf — Scarf specifically designed to facilitate mother-neonate skin-to-skin contact
  Arms: Scarf
Other: Usual clinical practice — Participants will receive the usual clinical practice
  Arms: Usual clinical practice

SUMMARY:
The skin-to-skin contact maneuver (kangaroo) has shown benefits in newborn babies. This is two-arm randomized open clinical trial to evaluate whether the use of a scarf specifically designed to facilitate the skin-to-skin method is effective in terms of increasing the skin-to-skin mother-neonate time, compared to traditional clinical practice. Mothers of full-term babies with expected delivery in the study centers will be included. Those mothers with a language barrier that prevents collaboration in the study procedures, cognitive impairment or morbid obesity will be excluded. The primary endpoint is the average daily skin-to-skin time during hospital admission days. A superiority analysis will be made in terms of the skin-to-skin time of the intervention arm, compared to the control arm.

ELIGIBILITY:
Inclusion Criteria:

- Moders attending the first hospital visit with the midwife, with delivery planned in either of the two study hospitals

Exclusion Criteria:

* Language barrier that prevents collaboration in the study procedures
* Cognitive impairment preventing collaboration in the study procedures
* Morbid obesity

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Enrollment: 143 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-21 (Actual)

PRIMARY OUTCOMES:
Mother-neonate skin-to-skin contact time (number of hours) | 72 hours
  Number of hours of skin-to-skin contact maneuver (kangaroo)

SECONDARY OUTCOMES:
Time in arms or in physical contact of the neonate with the mother / father | 72 hours
  Number of hours in arms or in physical contact of the neonate with the mother / father
Time of crying | 72 hours
  Number of hours crying
Newborn weight loss | 72 hours
  Weight change in grams
Parents satisfaction with hospital care | 72 hours
  Parents satisfaction (structured interview)

CONTACTS AND LOCATIONS:
Overall Officials: Marta Bernadó, Principal Investigator — Consorci Sanitari Alt Penedes i Garraf; Alejandro Rodríguez-Molinero, Study Director — Consorci Sanitari Alt Penedes i Garraf
Locations (1):
- Consorci Sanitari Alt Penedes i Garraf, Sant Pere de Ribes, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
IPD (without personal identification data) could be shared by requirement from other researchers after the end of the study, and only for research proposels and previous approval of promotor center of the study (CSAPG). Anyway, Spanish and European Union legal policy about data protection will strictly be followed (IPD will not be transferred outside European Union).
Supporting Information: Study Protocol, ICF
Time Frame: After publication of main results of the study
Access Criteria: IPD will be shared only for scientific research purposes and following the Spanish and European Union normative law about data protection. The requirements will be directed to the IP of the study. The IP will evaluate the request to verify and evaluate the data that is requested and the purposes for which it is requested. Next, the IP will transfer the request to the promotor center the study for the final decision.

REFERENCES:
- [Result] Bernado Vidal M, Galvez-Barron C, Perez-Lopez C, Adridar F, Mayol Fiol M, Ponce Molina MP, Herzog de Samaniego V, Saiz Sanz L, Miro B, Perez-Hoyos S, Torres Soto AJ, Martinez Dalmases R, Calero Bajoz T, Rodriguez-Molinero A. A specifically designed handkerchief for skin-to-skin care: A randomized controlled trial in Spain. Int J Gynaecol Obstet. 2025 Nov 11. doi: 10.1002/ijgo.70635. Online ahead of print. PMID 41216986